CLINICAL TRIAL: NCT05934500
Title: Effectiveness of Cannabidiol vs. Narcotics for Post Operative Pain Control in Elective Knee Arthroscopic Surgery
Brief Title: CBD Knee Scope Study
Acronym: CBDS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Foundation for Orthopaedic Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USF006030
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Opioid standard of care: Percocet (oxycodone 5mg-acetaminophen 325 mg) every 4 hours PRN postoperatively for 7 days
- Cannabidiol Oil 100 mg/day (Experimental): CDB 100mg PO liquid suspension QD starting 30 days prior to surgery and finishing 30 days post-operatively
  Interventions: Drug: Cannabidiol Oil
- Cannabidiol Oil 200 mg/day (Experimental): CBD 200mg PO liquid suspension QD starting 30 days prior to surgery and finishing 30 days post-operatively.
  Interventions: Drug: Cannabidiol Oil

INTERVENTIONS:
Drug: Cannabidiol Oil — Subjects will self administer CBD sublingually
  Arms: Cannabidiol Oil 100 mg/day; Cannabidiol Oil 200 mg/day

SUMMARY:
This is a prospective, randomized, nonblinded trial to evaluate the effectiveness of Cannabidiol (CBD) oil on post-operative pain control compared to opioid medications after a knee arthroscopy.

DETAILED DESCRIPTION:
This is a prospective non-blinded randomized controlled trial with 3 groups of subjects all undergoing knee arthroscopy for soft tissue pathology. The first group will receive the SOC opioid course: 7 days of Percocet (oxycodone 5mg-acetaminophen 325mg) every four hours PO PRN, following surgery. the second 100 mg CBD daily for 30 days pre-operatively continuing 30 days post-operatively, and the third group 200 mg CBD daily for 30 days pre-operatively continuing 30 days post-operatively.

All subjects in each of the three groups will undergo standard pre-operative and post-operative care, including physical exams, imaging, and education. They will only differ in pre-operative pain medication administration if they are in one of the two CBD groups. The groups will undergo surveys (sleep quality, self-reported pain, need for refill or switch to opioids). Sleep quality will be assessed with the Insomnia Severity Index (ISI) while pain, need for refill, and switch to opioids will be recorded by the patient on CRF packets. The CRF packets will be given to patients at each visit for them to fill out to the best of their ability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* requiring knee arthroscopy for soft tissue injury, acute or chronic knee injury
* able to complete surveys and follow-up visits

Exclusion Criteria:

* younger than 18 years of age
* history of knee dislocation, fracture, previous surgery, coexisting extremity pathology, *pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain control | 30 days post-operatively
  Numerical Pain Scale (NRS) 0 being no pain, 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Sleep Quality | 30 days preoperatively leading up to surgery, then 30 days postoperatively. Outcomes will be collected from surgery to 6 weeks postoperatively.
  Insomnia Severity Index .

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation for Orthopaedic Research and Education/ Florida Orthpaedic Institute, Tampa, Florida, United States